CLINICAL TRIAL: NCT04948827
Title: A Randomized, Double-Blind, Placebo-Controlled, First-In-Human Study to Assess Safety, Tolerability, and Pharmacokinetics of Single and Multiple Ascending Doses of SBP-9330 (With a Nested Food-Effect Arm) After Oral Administration in Healthy Subjects
Brief Title: A First-in-Human Study of SBP-9330 in Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Camino Pharma, LLC (Industry)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH); Sanford Burnham Prebys (Other); University of California, San Diego (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SBP-9330-101; U01DA051077 (NIH)
Record Dates: First submitted 2021-06-15; First posted 2021-07-02 (Actual); Results first posted 2024-04-16 (Actual); Last update posted 2024-04-16 (Actual); Status verified 2024-03

CONDITIONS: Smoking Cessation
MeSH Terms: conditions — Smoking Cessation

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (13):
- Part A1 - Single-Dose (Active; 150 mg ) (Experimental): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: SBP-9330
- Part A3 - Single-Dose Food Effect (Active; 225 mg) (Experimental): In this two-period food-effect cohort, each healthy nonsmoker subject received the randomly assigned treatment (SBP-9330 or placebo) under fasting conditions (Period 1). After a 7- to 14-day washout period, subjects received the same single dose of SBP-9330 or placebo in a fed state (Period 2) 30 minutes after the start of an FDA High-Fat and High-Calorie Breakfast. A sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: SBP-9330
- Part A2 - Single-Dose (Active; 300 mg) (Experimental): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: SBP-9330
- Part A4 - Single-Dose (Active; 450 mg) (Experimental): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: SBP-9330
- Part A5 - Single-Dose (Active; 600 mg) (Experimental): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: SBP-9330
- Part A - Single-Dose (Placebo; pooled) (Placebo Comparator): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects were randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Interventions: Drug: Placebo
- Part B1 - Multiple-Dose Active (150 mg) (Experimental): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: SBP-9330
- Part B2 - Multiple-Dose Active (225 mg) (Experimental): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: SBP-9330
- Part B3 - Multiple-Dose Active (300 mg) (Experimental): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: SBP-9330
- Part B - Multiple-Dose Placebo (pooled) (Placebo Comparator): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: Placebo
- Part C1 - Smoker Phase (Active; 150 mg) (Experimental): In Part C, cohorts of healthy smokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: SBP-9330
- Part C2 - Smoker Phase (Active; 225 mg) (Experimental): In Part C, cohorts of healthy smokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: SBP-9330
- Part C - Smoker Phase (Placebo; pooled) (Placebo Comparator): In Part C, cohorts of healthy smokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: SBP-9330 — SBP-9330 oral capsules
  Arms: Part A1 - Single-Dose (Active; 150 mg ); Part A2 - Single-Dose (Active; 300 mg); Part A3 - Single-Dose Food Effect (Active; 225 mg); Part A4 - Single-Dose (Active; 450 mg); Part A5 - Single-Dose (Active; 600 mg); Part B1 - Multiple-Dose Active (150 mg); Part B2 - Multiple-Dose Active (225 mg); Part B3 - Multiple-Dose Active (300 mg); Part C1 - Smoker Phase (Active; 150 mg); Part C2 - Smoker Phase (Active; 225 mg)
Drug: Placebo — Placebo oral capsules
  Arms: Part A - Single-Dose (Placebo; pooled); Part B - Multiple-Dose Placebo (pooled); Part C - Smoker Phase (Placebo; pooled)

SUMMARY:
This is a single center, first-in-human, randomized, double-blind, placebo-controlled, Single-Ascending Dose (SAD) / Multiple-Ascending Dose (MAD) study incorporating a food-effect cohort.

ELIGIBILITY:
Inclusion Criteria:

1. Provision of written informed consent prior to the initiation of any protocol-specific procedures
2. Stated willingness to comply with all study procedures and availability for the duration of the study
3. Healthy male or female subject ≥ 18 and ≤ 55 years of age
4. Body mass index (BMI) ≥ 18.5 kg/m2 and ≤ 32.0 kg/m2
5. Body weight ≥ 50.0 kg at Screening
6. A female subject must meet at least one of the following criteria: a. Is of childbearing potential and agrees to use an acceptable contraceptive method. b. Is of non-childbearing potential, defined as surgically sterile (i.e., has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation) or is in a postmenopausal state (i.e., at least 1 year without menses prior to the first study drug administration without an alternative medical condition and confirmed with a serum follicle-stimulating hormone [FSH] > 40 IU/L at Screening)
7. Male subjects, if not surgically sterilized, must agree to use adequate contraception and not donate sperm from the first admission to the CRU until 90 days after the last study drug administration.
8. Part A and B only: Never- or nonsmoker (a nonsmoker is defined as someone who completely stopped using nicotine products for at least 2 years prior to the first study drug administration)
9. Have no clinically significant medical or mental health conditions captured in the medical history or evidence of clinically significant findings on the physical examination and/or ECG, as determined by an Investigator
10. No clinically significant abnormalities in blood pressure, heart rate, body temperature and respiratory rate and no evidence of orthostatic hypotension or postural tachycardia at Screening.

    Part C Only:
11. Are current tobacco cigarette smokers who smoke an average of 10 or more cigarettes per day in the 30 days prior to Screening
12. Expired breath CO level ≥10 parts per million (ppm) at Screening and prior to the first study drug administration
13. Positive test result for cotinine at Screening and prior to the first study drug administration
14. Are not motivated to try to quit smoking from Screening through 30 days from the first study drug administration

Exclusion Criteria:

1. Female who is lactating
2. Female who is pregnant according to the pregnancy test at Screening or prior to the first study drug administration
3. Female who is planning to become pregnant during this study or within 90 days after the last study drug administration
4. Male with female partner who is pregnant, lactating, or planning to become pregnant during this study or within 90 days after the last study drug administration
5. Poor venous access as determined by an Investigator at Screening
6. History of significant hypersensitivity to SBP-9330 or any related products (including excipients of the formulations) as well as severe hypersensitivity reactions (like angioedema) to any drugs
7. Presence of any medical condition that, in the opinion of an Investigator, poses an unacceptable risk to the subjects
8. Presence or history of significant gastrointestinal, liver or kidney disease, or surgery that may affect drug absorption
9. Evidence or history of clinically significant cardiovascular, pulmonary, hematologic, psychiatric (including mood and substance use disorders), neurological (including migraines, seizures, and epilepsy), endocrine, renal, hepatic, gastrointestinal, immunologic or dermatologic disease
10. History of malignancy within the past five years, except for successfully treated basal cell carcinoma of the skin
11. History of suicidal ideation or suicidal behavior as per the C-SSRS questionnaire administered at Screening
12. Evidence or history of significant psychiatric disease or any DSM-5 disorder as assessed by the Mini International Neuropsychiatric Interview (M.I.N.I.) administered at Screening
13. Routine or chronic use of more than three grams of acetaminophen daily
14. Strenuous activity, sunbathing, and contact sports within 48 hours prior to (first) admission to the CRU
15. Current alcohol consumption exceeding two standard drinks per day on average (1 standard drink=10 grams of alcohol) for male subjects and one standard drink per day on average for female subjects
16. History of alcohol or drug (other than caffeine) use disorder within 12 months prior to Screening
17. Any clinically significant illness in the 28 days prior to the first study drug administration
18. QTcF interval (QT interval corrected for heart rate according to Fridericia) > 450 ms for males and > 470 ms for females at Screening or on Day -1
19. Parts A and B only: Positive test result for alcohol and/or drugs of abuse at Screening or prior to the first drug administration
20. Positive test results for HIV-1/HIV-2 antibodies, hepatitis B surface antigen or hepatitis C antibody
21. Consumption of any prescription drugs (with the exception of hormonal contraceptives or hormone replacement therapy) or over-the-counter medications and nutrients known to modulate cytochrome P450 (CYP450) enzymes activity (e.g., grapefruit or grapefruit juice, pomelo juice, star fruit, or Seville [blood] orange products) or St. John's Wort within 14 days prior to the first study drug administration
22. Consumption of other prescription and over-the-counter medication not specifically excluded by Exclusion Criterion 21 including health supplements and herbal remedies within 7 days prior to the first study drug administration (an exception is made for paracetamol [acetaminophen], which is allowed up to admission to the clinic).
23. Any other clinically significant abnormalities in laboratory test results at Screening that would, in the opinion of an Investigator, increase the subject's risk of participation, jeopardize complete participation in the study, or compromise interpretation of study data
24. Intake of an investigational product in the 30 days or 5 half-lives (whichever is longer) prior to Screening
25. Inclusion in a previous cohort of this clinical study
26. Employee of the contract research organization (CRO) or the Sponsor.
27. Blood donation (excluding plasma donation) of approximately 500 mL within 56 days prior to Screening
28. Plasma donation within 7 days prior to Screening

    Part C Only:
29. History of generalized rash reaction to any drugs
30. Positive test result (except cotinine) for alcohol and/or drugs of abuse at Screening or prior to the first study drug administration
31. Use of smoking cessation aids (NRT, bupropion, or varenicline) within 30 days prior to the first study drug administration
32. Unable to abstain from smoking tobacco cigarettes for at least 1 hour before and 2 hours after study drug administration
33. Unable to abstain from using nicotine-containing products other than tobacco cigarettes (e.g., pipes, cigars, e-cigarettes or vapes, nicotine topical patches, nicotine gum, or nicotine lozenges) during the study

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 90 (Actual)
Dates: Start 2021-07-20 (Actual); Primary Completion 2023-03-06 (Actual); Study Completion 2023-03-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Altasciences Clinical Kansas, Inc, Overland Park, Kansas, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- Part A1 Single Dose (Active; 150 mg); Part A2 - Single-Dose (Active; 300 mg); Part A4 - Single-Dose (Active; 450 mg); Part A5 - Single-Dose (Active; 600 mg); Part A - Single Dose - Placebo (Pooled): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
- Part A3 - Single-Dose Food-Effect (Active; 225 mg): In this two-period food-effect cohort, each healthy nonsmoker subject received the randomly assigned treatment (SBP-9330 or placebo) under fasting conditions (Period 1). After a 7- to 14-day washout period, subjects received the same single dose of SBP-9330 or placebo in a fed state (Period 2) 30 minutes after the start of an FDA High-Fat and High-Calorie Breakfast. A sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
- Part B1 - Multiple-Dose (Active; 150 mg); Part B2 - Multiple-Dose (Active; 225 mg); Part B3 - Multiple-Dose (Active; 300 mg); Part B - Multiple-Dose Placebo (Pooled): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
- Part C - Smoker Phase Placebo (Pooled): In Part C, cohorts of healthy smokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
Period: Overall Study
Arm/Group | Part A1 Single Dose (Active; 150 mg) | Part A3 - Single-Dose Food-Effect (Active; 225 mg) | Part A2 - Single-Dose (Active; 300 mg) | Part A4 - Single-Dose (Active; 450 mg) | Part A5 - Single-Dose (Active; 600 mg) | Part A - Single Dose - Placebo (Pooled) | Part B1 - Multiple-Dose (Active; 150 mg) | Part B2 - Multiple-Dose (Active; 225 mg) | Part B3 - Multiple-Dose (Active; 300 mg) | Part B - Multiple-Dose Placebo (Pooled) | Part C1 - Smoker Phase (Active; 150 mg) | Part C2 - Smoker Phase (Active; 225 mg) | Part C - Smoker Phase Placebo (Pooled)
Started | 6 | 6 | 6 | 6 | 6 | 10 | 8 | 8 | 8 | 6 | 8 | 8 | 4
Completed | 6 | 5 | 6 | 6 | 6 | 10 | 7 | 6 | 8 | 6 | 6 | 8 | 4
Not Completed | 0 | 1 | 0 | 0 | 0 | 0 | 1 | 2 | 0 | 0 | 2 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Part A1 - Single-Dose (Active; 150 mg ); Part A3 - Single-Dose (Active; 300 mg); Part A4 - Single-Dose (Active; 450 mg); Part A5 - Single-Dose (Active; 600 mg): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  SBP-9330: SBP-9330 oral capsules
- Part A2 - Single-Dose Food-Effect (Active; 225 mg): In this two-period food-effect cohort, each healthy nonsmoker subject received the randomly assigned treatment (SBP-9330 or placebo) under fasting conditions (Period 1). After a 7- to 14-day washout period, subjects received the same single dose of SBP-9330 or placebo in a fed state (Period 2) 30 minutes after the start of an FDA High-Fat and High-Calorie Breakfast. A sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  SBP-9330: SBP-9330 oral capsules
- Part A - Single Dose - Placebo (Pooled): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
  Placebo: Placebo oral capsules
- Part B1 - Multiple-Dose (Active; 150 mg); Part B2 - Multiple-Dose (Active; 225 mg); Part B3 - Multiple-Dose (Active; 300 mg): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  SBP-9330: SBP-9330 oral capsules
- Part C - Smoker Phase Placebo (Pooled): In Part C, cohorts of healthy smokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
  Placebo: Placebo oral capsules
- Total: Total of all reporting groups
Arm/Group | Part A1 - Single-Dose (Active; 150 mg ) | Part A2 - Single-Dose Food-Effect (Active; 225 mg) | Part A3 - Single-Dose (Active; 300 mg) | Part A4 - Single-Dose (Active; 450 mg) | Part A5 - Single-Dose (Active; 600 mg) | Part A - Single Dose - Placebo (Pooled) | Part B1 - Multiple-Dose (Active; 150 mg) | Part B2 - Multiple-Dose (Active; 225 mg) | Part B3 - Multiple-Dose (Active; 300 mg) | Part B - Multiple-Dose Placebo (Pooled) | Part C1 - Smoker Phase (Active; 150 mg) | Part C2 - Smoker Phase (Active; 225 mg) | Part C - Smoker Phase Placebo (Pooled) | Total
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 8 | 8 | 8 | 6 | 8 | 8 | 4 | 90
Age, Continuous [Mean (Standard Deviation); unit: years] | 30.5 (12.26) | 38.5 (10.09) | 35.3 (7.12) | 33.8 (9.41) | 32.2 (9.24) | 37.7 (11.44) | 34.0 (8.83) | 36.0 (8.57) | 38.5 (9.23) | 32.8 (11.69) | 40.3 (7.52) | 44.0 (8.28) | 39.8 (9.74) | 36.0 (9.24)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 5 | 3 | 4 | 0 | 3 | 3 | 5 | 3 | 3 | 0 | 2 | 3 | 2 | 36
  Male | 1 | 3 | 2 | 6 | 3 | 7 | 3 | 5 | 5 | 6 | 6 | 5 | 2 | 54
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 0 | 0 | 0 | 3 | 2 | 0 | 3 | 1 | 0 | 1 | 0 | 0 | 1 | 11
  Not Hispanic or Latino | 6 | 6 | 6 | 3 | 4 | 10 | 5 | 7 | 8 | 5 | 8 | 8 | 3 | 79
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Asian | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 2
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 1 | 0 | 0 | 1
  Black or African American | 3 | 4 | 4 | 3 | 4 | 4 | 2 | 4 | 1 | 3 | 3 | 1 | 2 | 38
  White | 3 | 2 | 2 | 3 | 1 | 6 | 4 | 4 | 6 | 3 | 2 | 7 | 2 | 45
  More than one race | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0 | 2 | 0 | 1 | 0 | 0 | 0 | 0 | 3
Region of Enrollment [Number; unit: participants]
  United States | 6 | 6 | 6 | 6 | 6 | 10 | 8 | 8 | 8 | 6 | 8 | 8 | 4 | 90
Body mass index [Mean (Standard Deviation); unit: kg/m^2] | 26.02 (4.005) | 28.70 (2.021) | 25.47 (3.755) | 28.97 (1.783) | 26.65 (2.643) | 26.20 (2.363) | 25.86 (2.529) | 27.38 (2.604) | 27.83 (3.290) | 25.13 (3.197) | 25.34 (4.489) | 26.98 (3.475) | 24.05 (3.884) | 26.2 (3.197)

OUTCOME MEASURES:

1. Primary Outcome: Number of Treatment-Emergent Adverse Events [Safety and Tolerability]
Description: Number of drug-related adverse events as determined by clinically significant changes in vital signs, physical examination findings, ECG parameters, C-SSRS questionnaire results, and clinical laboratory results
Time Frame: Part A: 8 days Part B: 21 days Part C: 21 days
Measure: Count of Participants; unit: Participants
Groups:
- A1 Single Dose (Active; 150 mg); Part A3 - Single-Dose (Active; 300 mg); Part A4 - Single-Dose (Active; 450 mg); Part A5 - Single-Dose (Active; 600 mg); Part A - Single Dose - Placebo (Pooled): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
- Part A2 - Single-Dose Food-Effect (Active; 225 mg): In this two-period food-effect cohort, each healthy nonsmoker subject received the randomly assigned treatment (SBP-9330 or placebo) under fasting conditions (Period 1). After a 7- to 14-day washout period, subjects received the same single dose of SBP-9330 or placebo in a fed state (Period 2) 30 minutes after the start of an FDA High-Fat and High-Calorie Breakfast. A sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data was completed prior to administration of doses to the remainder of the cohort.
- Active Comparator: Part B2 - Multiple-Dose (Active; 225 mg); Active Comparator: Part B3 - Multiple-Dose (Active; 300 mg); Part B - Multiple-Dose Placebo (Pooled): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
Arm/Group | A1 Single Dose (Active; 150 mg) | Part A2 - Single-Dose Food-Effect (Active; 225 mg) | Part A3 - Single-Dose (Active; 300 mg) | Part A4 - Single-Dose (Active; 450 mg) | Part A5 - Single-Dose (Active; 600 mg) | Part A - Single Dose - Placebo (Pooled) | Part B1 - Multiple-Dose (Active; 150 mg) | Active Comparator: Part B2 - Multiple-Dose (Active; 225 mg) | Active Comparator: Part B3 - Multiple-Dose (Active; 300 mg) | Part B - Multiple-Dose Placebo (Pooled) | Part C1 - Smoker Phase (Active; 150 mg) | Part C2 - Smoker Phase (Active; 225 mg) | Part C - Smoker Phase Placebo (Pooled)
Number analyzed (Participants) | 6 | 6 | 6 | 6 | 6 | 10 | 8 | 8 | 8 | 6 | 8 | 8 | 4
Participants | 0 | 1 | 1 | 1 | 1 | 2 | 7 | 4 | 5 | 4 | 4 | 7 | 1

2. Secondary Outcome: Pharmacokinetics of SBP-9330: Cmax
Description: Maximum observed concentration (Cmax)
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

3. Secondary Outcome: Pharmacokinetics of SBP-9330: Tmax
Description: Time to reach maximum observed concentration (Tmax)
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

4. Secondary Outcome: Pharmacokinetics of SBP-9330: AUC 0-24
Description: Area under the concentration time curve from time 0 (dose administration) to 24 hours
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 24 hours post-dose
Reporting Status: Not Posted

5. Secondary Outcome: Pharmacokinetics of SBP-9330: AUC 0-T
Description: Area under the concentration time curve from time 0 (dose administration) to the time of last quantifiable concentration
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

6. Secondary Outcome: Pharmacokinetics of SBP-9330: AUC 0-∞
Description: Area under the concentration time curve extrapolated to infinity
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

7. Secondary Outcome: Pharmacokinetics of SBP-9330: T½
Description: Terminal elimination half-life
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

8. Secondary Outcome: Pharmacokinetics of SBP-9330: CL/F
Description: Apparent total clearance
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

9. Secondary Outcome: Pharmacokinetics of SBP-9330: Vz/F
Description: Apparent volume of distribution
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

10. Secondary Outcome: Pharmacokinetics of SBP-9330: C Trough
Description: Observed concentration at the end of the dosing interval
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

11. Secondary Outcome: Pharmacokinetics of SBP-9330: Cτ
Description: Concentration at the end of the dosing interval.
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

12. Secondary Outcome: Pharmacokinetics of SBP-9330: AUCτ
Description: Area under the concentration time curve over the dosing interval at steady state, calculated from 0 to 24 hours (dosing interval)
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

13. Secondary Outcome: Pharmacokinetics of SBP-9330: T½, Eff
Description: Effective half-life
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

14. Secondary Outcome: Pharmacokinetics of SBP-9330: CL/Fss
Description: Apparent total clearance at steady state
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

15. Secondary Outcome: Pharmacokinetics of SBP-9330: Vz/Fss
Description: Apparent volume of distribution at steady state
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

16. Secondary Outcome: Pharmacokinetics of SBP-9330: RAC(Cmax)
Description: Accumulation ratio evaluated by comparing Day 14 Cmax to Day 1 Cmax
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

17. Secondary Outcome: Pharmacokinetics of SBP-9330: RAC(AUC)
Description: Accumulation ratio evaluated by comparing Day 14 AUCτ to Day 1 AUC0-24
Time Frame: PK samples were obtained at selected timepoints from pre-dose until 48 hours post-dose
Reporting Status: Not Posted

18. Other Pre Specified Outcome: Expired Carbon Monoxide (ECO) Level
Description: Expired breath CO was measured with a Bedfont Smokerlyzer™
Time Frame: Daily from Screening through Day 14
Reporting Status: Not Posted

19. Other Pre Specified Outcome: Plasma Cotinine Level
Description: Blood samples were collected to measure plasma cotinine levels
Time Frame: Predose, Day 7 and Day 14
Reporting Status: Not Posted

20. Other Pre Specified Outcome: Number of Cigarettes Smoked
Description: A daily smoking log was kept to document the number of cigarettes smoked
Time Frame: Daily from Screening through Day 14
Reporting Status: Not Posted

21. Other Pre Specified Outcome: Minnesota Nicotine Withdrawal Scale (MNWS)
Description: A self-report measure used to monitor symptoms of tobacco withdrawal.
Time Frame: Screening through Day 14
Reporting Status: Not Posted

22. Other Pre Specified Outcome: Questionnaire on Smoking Urges - Brief Version (QSU-Brief)
Description: A self-report questionnaire used to measure cravings to smoke.
Time Frame: Screening through Day 15
Reporting Status: Not Posted

ADVERSE EVENTS:
Time Frame: Part A: 8 days Part B: 21 days Part C: 21 days
Groups:
- Part A2 - Single-Dose (Active; 300 mg); Part A4 - Single-Dose (Active; 450 mg); Part A5 - Single-Dose (Active; 600 mg); Part A - Single Dose - Placebo (Pooled): In Part A, cohorts of healthy nonsmokers were randomized to either active SBP-9330 or matching placebo. In each cohort a sentinel group of 2 subjects was randomized and dosed ahead of the rest of the cohort. A review of safety data will be completed prior to administration of doses to the remainder of the cohort.
- Active Comparator: Part B3 - Multiple-Dose (Active; 225 mg); Active Comparator: Part B2 - Multiple-Dose (Active; 300 mg); Part B - Multiple-Dose Placebo (Pooled): In Part B, cohorts of healthy nonsmokers were randomized to receive once daily doses of active SBP-9330 or matching placebo for 14 consecutive days in increasing dose cohorts.
Arm/Group | A1 Single Dose (Active; 150 mg) | Part A3 - Single-Dose Food-Effect (Active; 225 mg) | Part A2 - Single-Dose (Active; 300 mg) | Part A4 - Single-Dose (Active; 450 mg) | Part A5 - Single-Dose (Active; 600 mg) | Part A - Single Dose - Placebo (Pooled) | Part B1 - Multiple-Dose (Active; 150 mg) | Active Comparator: Part B3 - Multiple-Dose (Active; 225 mg) | Active Comparator: Part B2 - Multiple-Dose (Active; 300 mg) | Part B - Multiple-Dose Placebo (Pooled) | Part C1 - Smoker Phase (Active; 150 mg) | Part C2 - Smoker Phase (Active; 225 mg) | Part C - Smoker Phase Placebo (Pooled)
All-Cause Mortality (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/4
Serious Adverse Events (participants affected / at risk) | 0/6 | 0/6 | 0/6 | 0/6 | 0/6 | 0/10 | 0/8 | 0/8 | 0/8 | 0/6 | 0/8 | 0/8 | 0/4
Other Adverse Events (participants affected / at risk) | 0/6 | 2/6 | 1/6 | 1/6 | 1/6 | 3/10 | 8/8 | 7/8 | 8/8 | 5/6 | 6/8 | 8/8 | 1/4
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | A1 Single Dose (Active; 150 mg) (N=6) | Part A3 - Single-Dose Food-Effect (Active; 225 mg) (N=6) | Part A2 - Single-Dose (Active; 300 mg) (N=6) | Part A4 - Single-Dose (Active; 450 mg) (N=6) | Part A5 - Single-Dose (Active; 600 mg) (N=6) | Part A - Single Dose - Placebo (Pooled) (N=10) | Part B1 - Multiple-Dose (Active; 150 mg) (N=8) | Active Comparator: Part B3 - Multiple-Dose (Active; 225 mg) (N=8) | Active Comparator: Part B2 - Multiple-Dose (Active; 300 mg) (N=8) | Part B - Multiple-Dose Placebo (Pooled) (N=6) | Part C1 - Smoker Phase (Active; 150 mg) (N=8) | Part C2 - Smoker Phase (Active; 225 mg) (N=8) | Part C - Smoker Phase Placebo (Pooled) (N=4)
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 2 (2) | 1 (1) | 1 (1) | 1 (1) | 2 (2) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 2 (2) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Presyncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Syncope (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Constipation (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 6 (6) | 1 (1)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flatulence (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal distention (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vomiting (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Orthostatic heart rate response increased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
White blood cell count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Neutrophil count decreased (Investigations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rhinorrhoea (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Dry throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Throat irritation (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Ecchymosis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Pruritus (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Chest discomfort (General disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Drug hypersensitivity (Immune system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
COVID-19 (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypochloraemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypokalemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hyponatremia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abnormal dreams (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Vaginal hemorrhage (Reproductive system and breast disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Abdominal discomfort (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Balance disorder (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Dyskinesia (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Insomnia (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Euphoric mood (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Ingrown hair (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Atrioventricular block second degree (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Influenza (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Epistaxis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Increased appetite (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Paresthesia oral (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2022-09-14): https://cdn.clinicaltrials.gov/large-docs/27/NCT04948827/Prot_000.pdf
  • Statistical Analysis Plan (2023-03-10): https://cdn.clinicaltrials.gov/large-docs/27/NCT04948827/SAP_001.pdf